CLINICAL TRIAL: NCT03345875
Title: Feasibility and Acceptability of HPV Self-Collection Cervical Cancer Screening and Treatment in Clinics and the Community in Botswana
Brief Title: Feasibility and Acceptability of HPV Self-Collection Cervical Cancer Screening and Treatment in Botswana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Botswana Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00007974
Record Dates: First submitted 2017-10-26; First posted 2017-11-17 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Human Papillomavirus Infection; Cervical Cancer
Keywords: human papillomavirus; cervical cancer; self-collection
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort study of women in an HPV self-collection screen-and-treat strategy for cervical cancer prevention to assess collection, triage and treatment through a service delivery model using descriptive, quantitative methods, and formative, qualitative research with providers and women.
  Methods to assess feasibility of the service model are electronic medical record (EMR) documentation of women's progression from eligibility for and receipt of services through each step of the HPV self-collection screen-and-treat strategy, from self-collection through test results to treatment of precancer, including referral for suspect cancer.
  Acceptability will entail: a) in-depth interviews with health providers, community mobilizers, health facility staff and managers and b) in-depth interviews and surveys with women who receive services as well as women that are eligible and decline services.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV Screening (Other): Study eligible participants will be screened for HPV using a self collected vaginal sample using a collection device and kit. Those who test positive for HPV will be offered visual assessment of the cervix for treatment (VAT) and treatment as appropriate.
  Interventions: Diagnostic Test: HPV self collection, followed by visual assessment of the cervix for treatment (VAT) and treatment

INTERVENTIONS:
Diagnostic Test: HPV self collection, followed by visual assessment of the cervix for treatment (VAT) and treatment — Women who test HPV positive are offered visual assessment for treatment, with treatment method (cryotherapy, LEEP, or biopsy) based on visual assessment findings.

SUMMARY:
Aims of the Study: To assess feasibility and acceptability of introducing HPV testing of self-collected vaginal specimens (self-collection for HPV) of women age 30-49 years, followed by visual assessment of the cervix for treatment (VAT) and treatment of women testing HPV positive at a district hospital, surrounding clinics and communities in Botswana.

Background and Rationale:

High HIV prevalence correlates with high rates of precancerous and cancerous changes on the cervix, and Botswana has the third highest HIV prevalence rate (22.2%) in the world. In Botswana, cervical cancer is the leading cause of cancer and cancer-related deaths among women. While the Government of Botswana has made cervical cancer a public health priority, and has provided cytology-based screening (Pap smears) for the past 20 years and in recent years began also offering VIA coupled with immediate cryotherapy for eligible precancerous lesions in a screen-and-treat (S&T) approach, the program still encounters multiple challenges. These include delays in reporting/receiving cytology results, referral bottlenecks for specialist care, and ultimately far fewer women being screened and treated than set targets. In response, in 2012 Botswana's Ministry of Health and Wellness (MoHW) developed a National Cervical Cancer Prevention Programme (NCCPP) Comprehensive Prevention and Control Strategy that includes implementing a demonstration project to gauge acceptability and obtain lessons that will be used in planning the roll-out of this screening method.

As a result, the MoHW is exploring human papillomavirus (HPV) testing as a primary screening method with the future service delivery in mind through HPV testing, specifically using self-collected samples, as a primary screening method. HPV testing is more sensitive and reliable for the detection of cervical precancer and cancer than Pap testing and VIA. This increased sensitivity translates into two important benefits: 1) earlier detection of significant precancerous lesions that if treated results in a ~50% reduction in the incidence of cervical cancer within 4-5 years compared to Pap testing and 50% reduction in related deaths within 8 years compared to Pap testing and VIA and 2) lower cancer risk for many years for those with a negative result, which permits screening at an extended interval of 5-10 years. The Xpert HPV test, which will be used in this study, has high sensitivity (100%) and relatively high specificity (81.5%) for CIN. HPV tests run on the GeneXpert® machine allow multiple tests (four in the model to be used in this study) to be run in an hour.

DETAILED DESCRIPTION:
A. Study Objectives:

Research Question 1. Is it feasible to implement HPV self-collection for cervical cancer prevention at a District Hospital, four surrounding clinics, and in the community among women eligible for cervical cancer screening per national guidelines, followed by VAT triage of HPV positive women at the clinic; and then treatment at the clinic or hospital?

* What is the HPV positivity rate (prevalence) for women age 30 - 49 years and disaggregated by HIV status and clinic location?
* What are the screening-to-treatment completion rates with this strategy for women with HPV-positive test, by HIV status and clinic location?

  * Can at least 75% of women doing HPV self-collection receive their results within 3 weeks self-collection?
  * Can at least 75% of women with an HPV positive result undergo VAT within 3 weeks of receiving their HPV result?
  * Can at least 90% of women with an HPV positive result undergo VAT and receive treatment within 3 months of initial HPV self-collection?

Research Question 2a, 2b. Do (2a) health care providers, community health workers, laboratory personnel, and managers and (2b) women consider the HPV self-collection, VAT and treatment acceptable? For each group of these participants, what are some of the enablers and the barriers to implementing an HPV self-collection screen-and-treat strategy?

B. Overview of Methods:

Research Question 1: Service Delivery Model The methods are prospective documentation of women's progression from eligibility for and receipt of services through each step of the HPV self-collection screen-and-treat strategy for cervical cancer prevention. This documentation and aggregation across client will involve client-level longitudinal data collected electronically from the time of HPV self-collection through test results to treatment of precancerous, including referral for suspect cancer cases as needed.

Research Question 2a and 2b:

Qualitative Research with Providers and Other Stakeholders:

The methods are in-depth interviews to be conducted with health providers, community mobilizers, health facility staff, and facility and district managers.

Mixed Method Research with Women: The methods are a combination of in-depth interviews and surveys to be conducted with women who receive services through each step of the HPV self-collection screen-and-treat strategy for cervical cancer prevention as well as women that are eligible and decline to do HPV self-collection.

C. Sample sizes and justifications by Research Question:

Hypothesis 1: Of eligible women who accept to do HPV self-collection, >75% will receive their HPV test results within 3 weeks. Summary from a statistical calculation: A sample size of 1022 women produces a two-sided 95% confidence interval with a width equal to 0.05 (5% precision on either side) when the sample proportion is 0.80

Research Question 1: Service Delivery Model

The study will include all women who meet eligibility criteria, consent and perform HPV self-collection up to 1,022 women. This will occur during a six-month enrollment period at the district hospital, four clinics or communities serviced by the clinics. By health facility, the break down is:

* Scottish Livingstone Hospital: 204 women
* Clinic 1: Lephephe: 103 women at the facility + 103 in the community
* Clinic 2: Thamaga 103 women at the facility + 103 in the community
* Clinic 3: Kopong: 203 women at the facility
* Clinic 4: Phuthadikobo: 203 women at the facility

Justification for Sample Size:

* The sample size of 1,022 is large enough to be meaningful to show the MoHW whether the HPV self-collection screen-and-treat strategy is feasible and acceptable.
* At any one time, up to 4 HPV tests can be run in the 1 GeneXpert machine dedicated for HPV tests, to be located at Scottish Livingstone Hospital. Processing takes 1 hour. Over 6 months, this is approximately 2 tests per working hour.
* The proportion of women who test HPV positive will result in the number of women to receive VAT and treatment.
* Based on historical data on women receiving treatment following VIA screening, we expect at least 85% of HPV-positive cases to be eligible for cryotherapy, which can be provided on the same day as the VAT. The sample size of 1,022 women will result in treatment services that are feasible to offer at Scottish Livingstone Hospital and Phuthadikobo Clinic.

Research Question 2a: Qualitative Research with Providers and Other Stakeholders.

In-depth interviews will be conducted at the district hospital and up to 4 clinics with the following persons: 2 VIA nurses, 1 doctor performing LEEP, 3 district management official, 6 facility or unit in-charges, 2 laboratory staff and 10 community mobilizers. Some participant types only work at district hospital while others are at the clinics. Up to 24 interviews will be conducted with providers and district authorities.

Research Question 2b: Qualitative and Survey Research with Women Among the women who do HPV self-collection, we will recruit clients from each facility or stated community, to participate in an in-depth interview. Among the women who test HPV positive and completes VAT, we will recruit two clients from each facility where the client is attached. Clients who fit the eligibility requirements, will be purposively recruited after completing her HPV self-collection, on a day when the interviewer is present at the facility in order to minimize burden and number of contacts with the client.

The qualitative sample size for questions 2a (24) and 2b (27) is a total of 51 interviews (Providers, Staff, Managers, and Clients). The sample size for RQ 2a is determined by the limited number of Providers, Staff, and Managers. The qualitative sample size for the number of women is determined to include women who may represent the variability of women's perceptions and experiences relevant to HPV self-testing and follow-up care to achieve saturation of themes.

D. Implementation In Research Question 1: Service Delivery Model, Step 1: Eligibility Assessment, Consent, Enrollment, and HPV Self-collection

* Health care worker informs and educates women attending clinics at SLH, at the Health Clinics, and in the community about cervical cancer, its prevention including HPV self-collection. Study staff recruit and screen women for eligibility for HPV self-collection at the facilities and this data is documented on the Eligibility Assessment Form, the Electronic Client Record 1 (ECR 1).
* Research nurse obtains informed consent of women who meet the study inclusion criteria and consent to HPV self-collection, and signature is collected within the Electronic Client Record as part of ECR 1.
* Research nurse collects basic demographic and contact information, including woman's telephone number(s) to allow for follow up with results. Research nurse asks the woman, and documents, if she prefers to be contacted with results by phone or in person at the facility.
* If HIV status is not known (no prior HIV testing or last documented HIV test result was negative but more than 12 months ago), research nurse recommends HIV testing and is excluded from the study until HIV status is documented by HIV testing and recorded on ECR 2.
* Research nurse provides HPV self-collection kit with a sampling brush (a broom-like device) and a PreservCyt solution vial to the woman and she is instructed on proper collection technique. The woman goes to a designated private area to self-collect the vaginal specimens and rinse the self-collection brush into the vial and caps the vial.
* The woman takes the vial of self-collected specimen to the research nurse who labels the specimen and records this information as well as the "ease of use" questions in the Electronic Client Record (ECR 2).

Step 2: Storage and transport of Self-collected specimens

* At hospital, self-collected specimens are HPV tested immediately, or, if not able to tested immediately that day, are stored at 2 - 30°C and tested later.
* In the community, study staff take the self-collected specimens to the study health clinic on the same day as collection.
* At the health clinic, the specimens are stored at 2 - 30°C.
* The specimens are transported at 2 - 30°C to SLH using the normal health clinic lab specimen transport mechanisms and schedule. Frequency of transport depends on the clinic, e.g., daily in some cases, but at least once a week

Step 3: HPV tests are run on GeneXpert® DX machine at hospital and results recorded in ECR

Step 4: The woman receives her HPV test results

* Senior Research Nurse or Research Assistant enters the HPV test of diagnosis into the electronic record data system (ECR 3), which can then be viewed by other study nurses at the study health clinic.
* Senior Research Nurse or Research Assistant notifies woman of HPV positivity/negativity in person or by phone, according to her preference, as noted in Step 1, and notification is documented in the ECR
* If the test is HPV positive, the woman is scheduled for a visit to a SLH VIA Clinic for VAT - possibly on same day.
* If the test is HPV negative, the woman is told her test is normal and should be retested in 3 year (HIV positive status) or 5 years (HIV negative status).

Step 5: VAT Note: Where VAT findings are eligible for cryotherapy, VAT (Step 5) and Treatment with cryotherapy (Step 6) mostly will occur during the same visit

• HPV-positive women will receive VAT. Nurses, midwives, and doctors, previously trained in VIA and cryotherapy, perform VAT and triage every client who is HPV-positive to determine treatment method and document findings in the electronic client record (ECR 4: VAT Result and ECR 6: Referral Result).

Possible VIA findings:

* VIA-negative (no lesion seen) - eligible for cryotherapy
* VIA-positive - eligible for cryotherapy: not suspicious for cancer, small lesion (meets standard eligibility criteria for cryotherapy); or
* VIA-positive - not eligible for cryotherapy: Large lesion, not eligible for cryotherapy, referred to the LEEP Clinic at SLH; or
* Suspicious for cancer: referred to Colposcopy/LEEP Clinic at SLH for further management.

Step 6: Treatment

* Following VAT, women eligible for cryotherapy are offered immediate treatment and treatment is performed according to standards. Treatment is documented in the electronic client record (ECR 4: VAT Result).
* Following VAT, women with large lesions are referred to the SLH LEEP Clinic, where LEEP is performed according to standards. Treatment is documented in the electronic client record (ECR 6: Referral Result and ECR 4: VAT Result).
* Following VAT, women with suspect cancer are referred to the SLH Colposcopy/LEEP Clinic, where biopsies are obtained and further management is arranged. Management is documented in the electronic client record (ECR 6: Referral Result).
* Following treatment, healthcare worker counsels the woman on findings, self-care, and warning signs and to return in one year for rescreening

In Research Question 2a, the qualitative interviewer will meet with the consenting provider or other stakeholder in a private room. The interview will cover the experiences and opinions of providers, staff and managers on the various features in using the HPV test and self-collection, and other implementation considerations such as impact of the program on the quality of services and potential uptake within the community. These interviews will be conducted towards the end of the 6 month implementation period, to allow for participants to develop opinions and fully answer questions related to sustainability. Interviews with providers, community mobilizers, stakeholders and other Ministry employees will be conducted in English or Setswana, depending on the participant preference, and last up to an hour in length.

In Research Question 2b, in a private room, the qualitative interviewer will meet with consenting women who accept HPV self-collection and with consenting women who are HPV positive and return for VAT. The Senior Research Nurse or Research Assistant will meet with consenting women in a private to conduct surveys on women who are eligible but do not accept to do HPV self-collection, and women who are HPV positive but do not return for VAT within two weeks of receiving their results. Surveys will assess their reasons for not accepting self-testing for HPV or not returning for VAT. Interviews and Surveys under Research Question 2b will be fit into the same Service Delivery Model previously described.

E. Data Analysis Data analysis will be descriptive with no statistical testing planned since the research questions are descriptive. We will report confidence intervals around mean values of indicators, also median and interquartile range, when appropriate.

Qualitative data will be transcribed, and translated. Analysts will come up with an initial codebook, a list of draft codes based on our field guide questions and anticipating some themes and sub-themes from reading the literature.

Each transcript will be coded and considered for analysis in the same way. We will allow for and encourage addition of emergent codes. Once we code all transcripts, we will divide up the codes into code families. After reading through passages in a code family, we will create a display matrix following the framework analysis approach. In this display, each participant is a row and each theme and sub-theme is a column, cells refer to specific quotes; this will allow for comparisons of the narratives among different types of participants. This visual matrix allows the analyst to move back and forth between different levels of abstraction and facilitates cross-case and within-case analyses.

The final phase of analysis, abstraction and interpretation will follow these steps: a) categorization, in which the researcher takes note of, and may write memos to document, the range and diversity of views, underlying dimensions of themes and creates categories; b) mapping linkages and connections and allowing for creation of typologies; and c) explanation, which involves accounting for the patterns of association in the data, and considering alternative explanations.

F. Protection of participants Clients' non-participation in any aspect of the study or withdrawal from our study will NOT affect their health care or their employment. Information that we gain from the quantitative, qualitative, or analysis components will not be shared with any individual or organization (i.e. government authorities, NGO representatives) except in aggregate form, and the results will have no participant identifiers.

A separate database that links the national ID numbers/passport number and client's name the unique study ID numbers will be kept in a separate password protected, electronic database that only study staff will be able to access. Study team members will clearly explain the purpose of the study to the facility representatives and other participants, as well as obtain written informed consent from participants for participation in the service delivery process and in the qualitative interviews. Data collectors will be trained to be sensitive and to answer any questions. A strategy for keeping data confidential will be developed and followed.

All individual recruitment of any woman or provider participant will occur in a space at the facility, or community, that allows for audio and visual privacy (not in open view or in a place where others can overhear the conversation). The research nurse will be trained to seek a private space for the recruitment To ensure that the data will be kept confidential and secure, data collection team/interviewers will be trained on issues of ethics and will sign confidentiality agreements to ensure that they do not share the completed data collection tools outside study team. The completed notes from interviews and will be sealed in envelopes immediately after the completion of data collection. Electronically entered data will be password protected upon entry. Paper-based and electronic data, including audio files, will be kept safe in locked containers and transported to the Jhpiego offices in Gaborone. Audio files and transcripts of the de-identified key informant interviews will be stored in a password protected, compressed folder, which will be upload to a password-protected Dropbox folder, a web-based software application to share files with data analysts at Jhpiego Botswana and Baltimore. Hard copies of data will be kept in locked cupboards. The data will be entered in an electronic database accessible only to authorized assessment personnel.

G. Risks or Discomforts to Participants HPV test self-collection is the main focus of the investigation in this study. This study will use the standard of care treatments available in Botswana for women who test HPV positive. The VIA used in VAT and treatment are not under investigation. We do not foresee adverse events. It is possible that there could be misunderstandings about the HPV self-collection at the community level; therefore we will make sure that community leaders and members are sensitized to the purpose and procedures of the study at the facility and community level.

An adverse event would be considered a disclosure of client information due to the study. As precautions will be taken to protect client information with confidentiality (as described above), adverse events are unlikely. The study team will follow up on each enrolled participant's case to make sure each woman has received services. If we learn of any adverse event with an enrolled participant, we will follow up to learn the nature of the problem.

The PI, Dr. John Varallo, Jhpiego, will be in constant communication with the Jhpiego-Botswana Country Team on the progress of the study and will contact the MOHW and the JHSPH IRB in case of any problems. They will try to quickly resolve any problems that arise.

ELIGIBILITY:
The District Health Management Team (DHMT), estimates that in 2011 there were 31,574 women 30-49 years of age on the Kweneng East catchment area, serviced by Scottish Livingstone Hospital and the 4 selected Health Clinics.

Women will be clients of the health facility at one of the clinics (described below under recruitment), may come to the facility for cervical cancer screening after having been contacted by a community mobilizer, or women attending a community health campaign event (in the community).

Participants under Research Question 1: 1022 women Participants under Research Question 2a: 24 providers and other stakeholders Participants under Research Question 2b: 27 women for in-depth interviews; 250 women for structured surveys.

Inclusion Criteria: Service Delivery Model

* Age 30 to 49 years,
* Not screened recently/never screened before, defined as:

  * No prior history of cervical cancer screening: Pap smear, VIA or HPV testing), or
  * Prior screening, but result unknown and no treatment
  * Prior screening occurred more than 5 years ago for HIV negative women or 3 years ago for HIV positive women
* HIV status is known (HIV positive result, or documented HIV negative result is less than 12 months ago).
* No history of prior abnormal screening or treatment/procedure on her cervix due to abnormal screening
* No history of cervical cancer
* Not currently pregnant; not less than 6 weeks postpartum
* Intact uterus/ no prior hysterectomy with a cervix present
* Accesses services in Kweneng East District study catchment area
* Able and willing to provide consent

Inclusion Criteria: Qualitative Research with Providers and Other Stakeholders

* Working as one of the cadres in Sampling Table 1 at the time of the interview.
* Working in cervical cancer prevention currently.
* Manager agrees the participant can take part in interview.
* Has been trained by the study regarding HPV self-collection and VAT.
* Willing to participate in in-depth interview and gives informed consent.

Exclusion Criteria:

* Woman does not meet the criteria for inclusion age 29 years or younger and age 50 years or older.
* Screened for cervical cancer in last 3 years if HIV positive, or in the last 5 years if HIV negative.
* Had an abnormal cervical cancer screening and/ or treatment of cervix ,
* History of cervical cancer HIV status unknown,
* Pregnant (self-report or by pregnancy test confirmation.
* Less than 6 weeks postpartum, prior hysterectomy,
* Unable to participate and give informed consent.
* Not interested in HPV self-collection.
* Unwilling to give informed consent

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 1022 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Screening-to-treatment completion rates for assessing feasibility of HPV self collection, VAT screening and treatment | 3 months per participant
  This outcome will be assessed by: the screening-to-treatment completion rates with this strategy for women with HPV-positive test, by HIV status and clinic location;
Qualitative interviews and surveys to assess acceptability of HPV Self Collection from women | At time of return for VAT for women who are HPV positive; At the time of declining VAT for women who are HPV positive; At the time of decline to self collect at all.
  Qualitative interview field guides and surveys will be given to elicit opinions from women on the acceptability and feasibility of using HPV self-collection and VAT at the facility and community-level
Qualitative interviews and surveys to assess acceptability of HPV Self Collection from health providers and managers | 6 months after the intervention has started at each facility, with a sampling of types of personnel
  Qualitative interview field guides and surveys will be given to elicit opinions from providers, staff, managers, community health workers, laboratory personnel on the acceptability and feasibility of using HPV in their facilities including self-collection, VAT and treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Varallo, MD, Principal Investigator — Jhpiego
Locations (5):
- Botswana (5):
  - Kopong Health Clinic, Kopong
  - Lephepe Health Clinic, Lephepe
  - Phuthadikobo, Molepolole
  - Scottish Livingstone Hospital, Molepolole
  - Thamaga Health Clinic, Thamaga

REFERENCES:
- [Background] WHO Guidelines for Screening and Treatment of Precancerous Lesions for Cervical Cancer Prevention. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK195239/ PMID 24716265
- [Background] UNAIDS. "AIDSinfo." At: http://aidsinfo.unaids.org/. Accessed 11 November 2016
- [Background] Botswana, Ministry of Health, "Five-year Comprehensive Prevention and Control Strategy (2012 - 2016)"
- [Background] Cuzick J, Clavel C, Petry KU, Meijer CJ, Hoyer H, Ratnam S, Szarewski A, Birembaut P, Kulasingam S, Sasieni P, Iftner T. Overview of the European and North American studies on HPV testing in primary cervical cancer screening. Int J Cancer. 2006 Sep 1;119(5):1095-101. doi: 10.1002/ijc.21955. PMID 16586444
- [Background] Mayrand MH, Duarte-Franco E, Rodrigues I, Walter SD, Hanley J, Ferenczy A, Ratnam S, Coutlee F, Franco EL; Canadian Cervical Cancer Screening Trial Study Group. Human papillomavirus DNA versus Papanicolaou screening tests for cervical cancer. N Engl J Med. 2007 Oct 18;357(16):1579-88. doi: 10.1056/NEJMoa071430. PMID 17942871
- [Background] Naucler P, Ryd W, Tornberg S, Strand A, Wadell G, Elfgren K, Radberg T, Strander B, Johansson B, Forslund O, Hansson BG, Rylander E, Dillner J. Human papillomavirus and Papanicolaou tests to screen for cervical cancer. N Engl J Med. 2007 Oct 18;357(16):1589-97. doi: 10.1056/NEJMoa073204. PMID 17942872
- [Background] Rijkaart DC, Berkhof J, Rozendaal L, van Kemenade FJ, Bulkmans NW, Heideman DA, Kenter GG, Cuzick J, Snijders PJ, Meijer CJ. Human papillomavirus testing for the detection of high-grade cervical intraepithelial neoplasia and cancer: final results of the POBASCAM randomised controlled trial. Lancet Oncol. 2012 Jan;13(1):78-88. doi: 10.1016/S1470-2045(11)70296-0. Epub 2011 Dec 14. PMID 22177579
- [Background] Ronco G, Giorgi-Rossi P, Carozzi F, Confortini M, Dalla Palma P, Del Mistro A, Ghiringhello B, Girlando S, Gillio-Tos A, De Marco L, Naldoni C, Pierotti P, Rizzolo R, Schincaglia P, Zorzi M, Zappa M, Segnan N, Cuzick J; New Technologies for Cervical Cancer screening (NTCC) Working Group. Efficacy of human papillomavirus testing for the detection of invasive cervical cancers and cervical intraepithelial neoplasia: a randomised controlled trial. Lancet Oncol. 2010 Mar;11(3):249-57. doi: 10.1016/S1470-2045(09)70360-2. Epub 2010 Jan 18. PMID 20089449
- [Background] Castle PE, Stoler MH, Wright TC Jr, Sharma A, Wright TL, Behrens CM. Performance of carcinogenic human papillomavirus (HPV) testing and HPV16 or HPV18 genotyping for cervical cancer screening of women aged 25 years and older: a subanalysis of the ATHENA study. Lancet Oncol. 2011 Sep;12(9):880-90. doi: 10.1016/S1470-2045(11)70188-7. Epub 2011 Aug 22. PMID 21865084
- [Background] Castle PE, Wheeler CM, Solomon D, Schiffman M, Peyton CL; ALTS Group. Interlaboratory reliability of Hybrid Capture 2. Am J Clin Pathol. 2004 Aug;122(2):238-45. doi: 10.1309/BA43-HMCA-J26V-WQH3. PMID 15323141
- [Background] Carozzi FM, Del Mistro A, Confortini M, Sani C, Puliti D, Trevisan R, De Marco L, Tos AG, Girlando S, Palma PD, Pellegrini A, Schiboni ML, Crucitti P, Pierotti P, Vignato A, Ronco G. Reproducibility of HPV DNA Testing by Hybrid Capture 2 in a Screening Setting. Am J Clin Pathol. 2005 Nov;124(5):716-21. doi: 10.1309/84E5-WHJQ-HK83-BGQD. PMID 16203283
- [Background] Stoler MH, Schiffman M; Atypical Squamous Cells of Undetermined Significance-Low-grade Squamous Intraepithelial Lesion Triage Study (ALTS) Group. Interobserver reproducibility of cervical cytologic and histologic interpretations: realistic estimates from the ASCUS-LSIL Triage Study. JAMA. 2001 Mar 21;285(11):1500-5. doi: 10.1001/jama.285.11.1500. PMID 11255427
- [Background] Ronco G, Dillner J, Elfstrom KM, Tunesi S, Snijders PJ, Arbyn M, Kitchener H, Segnan N, Gilham C, Giorgi-Rossi P, Berkhof J, Peto J, Meijer CJ; International HPV screening working group. Efficacy of HPV-based screening for prevention of invasive cervical cancer: follow-up of four European randomised controlled trials. Lancet. 2014 Feb 8;383(9916):524-32. doi: 10.1016/S0140-6736(13)62218-7. Epub 2013 Nov 3. PMID 24192252
- [Background] Sankaranarayanan R, Nene BM, Shastri SS, Jayant K, Muwonge R, Budukh AM, Hingmire S, Malvi SG, Thorat R, Kothari A, Chinoy R, Kelkar R, Kane S, Desai S, Keskar VR, Rajeshwarkar R, Panse N, Dinshaw KA. HPV screening for cervical cancer in rural India. N Engl J Med. 2009 Apr 2;360(14):1385-94. doi: 10.1056/NEJMoa0808516. PMID 19339719
- [Background] Dillner J, Rebolj M, Birembaut P, Petry KU, Szarewski A, Munk C, de Sanjose S, Naucler P, Lloveras B, Kjaer S, Cuzick J, van Ballegooijen M, Clavel C, Iftner T; Joint European Cohort Study. Long term predictive values of cytology and human papillomavirus testing in cervical cancer screening: joint European cohort study. BMJ. 2008 Oct 13;337:a1754. doi: 10.1136/bmj.a1754. PMID 18852164
- [Background] Castle PE, Glass AG, Rush BB, Scott DR, Wentzensen N, Gage JC, Buckland J, Rydzak G, Lorincz AT, Wacholder S. Clinical human papillomavirus detection forecasts cervical cancer risk in women over 18 years of follow-up. J Clin Oncol. 2012 Sep 1;30(25):3044-50. doi: 10.1200/JCO.2011.38.8389. Epub 2012 Jul 30. PMID 22851570
- [Background] Katki HA, Kinney WK, Fetterman B, Lorey T, Poitras NE, Cheung L, Demuth F, Schiffman M, Wacholder S, Castle PE. Cervical cancer risk for women undergoing concurrent testing for human papillomavirus and cervical cytology: a population-based study in routine clinical practice. Lancet Oncol. 2011 Jul;12(7):663-72. doi: 10.1016/S1470-2045(11)70145-0. Epub 2011 Jun 16. PMID 21684207
- [Background] Integrating HPV testing in cervical cancer screening program: a manual for program managers. Washington, D.C.: PAHO, 2016.
- See also: UNAIDS Accessed 11 November 2016 — http://aidsinfo.unaids.org/
- See also: 2014 Botswana AIDS Response Progress Report — http://www.unaids.org/en/regionscountries/countries/botswana
- See also: GLOBOCAN 2012. Population Factsheet. Accessed 10 November 2016 — http://globocan.iarc.fr